CLINICAL TRIAL: NCT05059561
Title: Temperament and Character Traits in Young Men Diagnosed With Idiopathic Scoliosis
Brief Title: Temperament and Character Traits in Young Men With Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Ozgur Maden, PhD. MD., Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: Sultan Abdulhamid TRH
Record Dates: First submitted 2021-09-19; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Idiopathic Scoliosis
Keywords: Idiopathic scoliosis; temperament; character; personality; persistence; novelty-seeking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients group: All patients who applied to the orthopedics and traumatology department between July 2017 and June 2018 for a medical board examination were evaluated by physical and radiological examination. According to the Cobb method, individuals with a Cobb angle greater than 10° were diagnosed with Idiopathic Scoliosis. All participants were evaluated by a senior psychiatrist. Before the interview, all subjects fully informed about the purpose and scope of the study. After their permission was obtained the study and control groups completed a socio-demographic data form consisting of questions about detailed personal and medical history and, the participants were asked to fill in the TCI.
  Interventions: Radiation: X-ray radiograghy
- Control group: All patients who applied to the orthopedics and traumatology department between July 2017 and June 2018 for a medical board examination were evaluated by physical and radiological examination. Healthy individuals who applied for the same examination and met the inclusion criteria were determined as the control group by random sampling method. All participants were evaluated by a senior psychiatrist. Before the interview, all subjects fully informed about the purpose and scope of the study. After their permission was obtained the control group completed a socio-demographic data form consisting of questions about detailed personal and medical history and, the participants were asked to fill in the TCI.
  Interventions: Radiation: X-ray radiograghy

INTERVENTIONS:
Radiation: X-ray radiograghy — Cobb angles of the patient and control groups were determined by using X-Ray radiography used in the radiological examination routinely applied to the individuals who applied for the health board examination.

SUMMARY:
This study was designed to investigate whether the temperament and character traits of young men with idiopathic scoliosis differ from healthy individuals of the same age group and characteristics.

DETAILED DESCRIPTION:
All patients who applied to the orthopedics and traumatology department between July 2017 and June 2018 for a medical board examination were evaluated by physical and radiological examination. According to the Cobb method, individuals with a Cobb angle greater than 10° were diagnosed with Idiopathic Scoliosis. In the same period, healthy individuals who applied for the same examination and met the inclusion criteria were determined as the control group by random sampling method. All participants were evaluated by a senior psychiatrist. Before the interview, all subjects fully informed about the purpose and scope of the study. After their permission was obtained the study and control groups completed a socio-demographic data form consisting of questions about detailed personal and medical history and, the participants were asked to fill in the TCI.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were 18 years of age and older, adequate level of education (at least primary school graduates) and capable of taking the tests and structured interview form, agreed to participate in the study, diagnosed with IS and did not have any psychiatric follow-up and treatment history.

Exclusion Criteria:

Individuals who were younger than 18 years of age, did not accept to participate in the study, had psychiatric disorders according to DSM V diagnostic criteria, additional medical disorders, and who were not at the level of education to take the tests and structured interview form were excluded from the study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Young men over 18 years of age were included in the study.
Study Population: Patient group: 162 person Control group: 162 person
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Temperament and Character Traits in Young Men Diagnosed With Idiopathic Scoliosis - First Evaluation | July 2017-July 2018
  Examining the X-ray radiograph results of all individuals who applied for a medical board examination report between July 2017 and July 2018, and identifying those with and without idiopathic scoliosis

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Abdulhamid Han Training and Research Hospital, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If requested, the study data can be accessed when deemed appropriate by the authors, provided that the identity information of the participants is kept confidential.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: There is no timeframe.

REFERENCES:
- [Background] Kuloğlu M, Sağlam S, Korkmaz S et. al. Temperament and character traits and alexithymia in patients with multiple sclerosis. Archives of Neuropsychiatry, 2013;50(1):34-40.
- [Background] Lundberg G, Anderberg UM, Gerdle B. Personality features in female fibromyalgia syndrome. J Musculosketal Pain, 2009;17: 117-130.
- [Result] Arnett JJ. Emerging adulthood. A theory of development from the late teens through the twenties. Am Psychol. 2000 May;55(5):469-80. PMID 10842426
- [Result] Cloninger CR, Svrakic DM, Przybeck TR. A psychobiological model of temperament and character. Arch Gen Psychiatry. 1993 Dec;50(12):975-90. doi: 10.1001/archpsyc.1993.01820240059008. PMID 8250684
- [Result] Cloninger CR. Temperament and personality. Curr Opin Neurobiol. 1994 Apr;4(2):266-73. doi: 10.1016/0959-4388(94)90083-3. PMID 8038587
- [Result] Cobb JR. Outline for the study of scoliosis. American Academy of Orthopaedic Surgeons Instructional Course Lectures, 1948;5: 261-265.
- [Result] Fadzan M, Bettany-Saltikov J. Etiological Theories of Adolescent Idiopathic Scoliosis: Past and Present. Open Orthop J. 2017 Dec 29;11:1466-1489. doi: 10.2174/1874325001711011466. eCollection 2017. PMID 29399224
- [Result] Fisher S, Cleveland SE. Body image and personality. Princeton, NJ: Nostrand, 1958.
- [Result] Freidel K. Psychosocial problems in idiopathic scoliosis. Retrieved from: Berlin: dissertation.de, 1999.
- [Result] Gokmen F, Altinbas K, Akbal A, Celik M, Savas Y, Gokmen E, Resorlu H, Karaca A. Evaluation of the temperament and character properties of patients with ankylosing spondylitis. Z Rheumatol. 2014 Nov;73(9):843-7. doi: 10.1007/s00393-013-1336-1. PMID 24549924
- [Result] Grauers A, Einarsdottir E, Gerdhem P. Genetics and pathogenesis of idiopathic scoliosis. Scoliosis Spinal Disord. 2016 Nov 28;11:45. doi: 10.1186/s13013-016-0105-8. eCollection 2016. PMID 27933320
- [Result] Grucza RA, Przybeck TR, Cloninger CR. Prevalence and correlates of binge eating disorder in a community sample. Compr Psychiatry. 2007 Mar-Apr;48(2):124-31. doi: 10.1016/j.comppsych.2006.08.002. Epub 2006 Nov 9. PMID 17292702
- [Result] Hresko MT, Talwalkar V, Schwend R; AAOS, SRS, and POSNA. Early Detection of Idiopathic Scoliosis in Adolescents. J Bone Joint Surg Am. 2016 Aug 17;98(16):e67. doi: 10.2106/JBJS.16.00224. No abstract available. PMID 27535448
- [Result] Kasai Y, Takegami K, Uchida A. A study of patients with spinal disease using Maudsley Personality Inventory. Int Orthop. 2004 Feb;28(1):56-9. doi: 10.1007/s00264-003-0489-y. Epub 2003 Jul 8. PMID 12851787
- [Result] Konieczny MR, Senyurt H, Krauspe R. Epidemiology of adolescent idiopathic scoliosis. J Child Orthop. 2013 Feb;7(1):3-9. doi: 10.1007/s11832-012-0457-4. Epub 2012 Dec 11. PMID 24432052
- [Result] Köse S, Sayar K, Ak İ et. al. Temperament and Character Inventory (Turkish TCI): Validity, reliability and factor structure. Bulletin of Clinical Psychopharmacology, 2004;14: 107-131.
- [Result] Mancuso SG, Knoesen NP, Chamberlain JA et. al. The temperament and character profile of a body dysmorphic disorder outpatient sample. Personality and Mental Health, 2009;3(4): 284-294.
- [Result] Misterska E, Glowacki M, Harasymczuk J. Personality characteristics of females with adolescent idiopathic scoliosis after brace or surgical treatment compared to healthy controls. Med Sci Monit. 2010 Dec;16(12):CR606-15. PMID 21119579
- [Result] Oh CH, Shim YS, Yoon SH, Park HC, Park CO, Lee MS. The psychopathological influence of adolescent idiopathic scoliosis in korean male : an analysis of multiphasic personal inventory test results. J Korean Neurosurg Soc. 2013 Jan;53(1):13-8. doi: 10.3340/jkns.2013.53.1.13. Epub 2013 Jan 31. PMID 23440382
- [Result] Özgüven İE. University students' problems and ways of coping. Hacettepe University Journal of Faculty of Education, 1992;7(7):5-13.
- [Result] Pyatakova GV, Okoneshnikova OV, Kozhevnikova AO et. al. Psychological aspects of treatment and rehabilitation of patients with adolescent idiopathic scoliosis: Research analysis. Pediatric Traumatology, Orthopaedics and Reconstructive Surgery, 2019;7(2):103-115.
- [Result] Saccomani L, Vercellino F, Rizzo P, Becchetti S. [Adolescents with scoliosis: psychological and psychopathological aspects]. Minerva Pediatr. 1998 Jan-Feb;50(1-2):9-14. Italian. PMID 9658793
- [Result] Schatzinger LH, Brower EM, Nash CL Jr. The patient with scoliosis. Spinal fusion: emotional stress and adjustment. Am J Nurs. 1979 Sep;79(9):1608-12. No abstract available. PMID 258574
- [Result] Smith FM, Latchford G, Hall RM, Millner PA, Dickson RA. Indications of disordered eating behaviour in adolescent patients with idiopathic scoliosis. J Bone Joint Surg Br. 2002 Apr;84(3):392-4. doi: 10.1302/0301-620x.84b3.12619. PMID 12002499
- [Result] Sullivan S, Cloninger CR, Przybeck TR, Klein S. Personality characteristics in obesity and relationship with successful weight loss. Int J Obes (Lond). 2007 Apr;31(4):669-74. doi: 10.1038/sj.ijo.0803464. Epub 2006 Sep 5. PMID 16953251
- [Result] Weinstein SL, Dolan LA, Spratt KF, Peterson KK, Spoonamore MJ, Ponseti IV. Health and function of patients with untreated idiopathic scoliosis: a 50-year natural history study. JAMA. 2003 Feb 5;289(5):559-67. doi: 10.1001/jama.289.5.559. PMID 12578488
- [Result] Weinstein SL. The Natural History of Adolescent Idiopathic Scoliosis. J Pediatr Orthop. 2019 Jul;39(Issue 6, Supplement 1 Suppl 1):S44-S46. doi: 10.1097/BPO.0000000000001350. PMID 31169647
- [Result] Weiss HR, Lehnert-Schroth C, Moramarco M. Schroth therapy: Advancements in conservative scoliosis treatment. Moldova, LAP Lambert Academic Publishing, 2018.
- [Result] Yilmaz H, Zateri C, Kusvuran Ozkan A, Kayalar G, Berk H. Prevalence of adolescent idiopathic scoliosis in Turkey: an epidemiological study. Spine J. 2020 Jun;20(6):947-955. doi: 10.1016/j.spinee.2020.01.008. Epub 2020 Jan 20. PMID 31972303